CLINICAL TRIAL: NCT03025607
Title: A Mixed Methods Pilot Randomized Controlled Trial of a Mobile Phone-based Health Program Among Adults With Prediabetes
Brief Title: A Mobile Phone-based Program for Adults With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Mary Ellen Michele Heisler, Dr. Michele Heisler, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2420.PIRAP
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Prediabetic State; Diabetes Mellitus
Keywords: Prevention; Mobile health; Autonomous motivation
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in this group will receive information on prediabetes and evidence-based ways to decrease progression to diabetes as well as a list of resources for mHealth tools for monitoring diet, physical activity, and weight.
- JOOL-Only (Experimental): Participants in this group will receive information on prediabetes and evidence-based ways to decrease progression to diabetes, a list of resources for mHealth tools to monitor diet, physical activity and weight, and will receive the JOOL Health mobile phone application.
  Interventions: Device: JOOL Health Mobile Phone Application
- JOOL-Plus (Experimental): Participants in this group will receive information on prediabetes and evidence-based ways to decrease progression to diabetes, a list of resources for mHealth tools to monitor diet, physical activity and weight, the JOOL Health mobile phone application, a digital scale, and a Fitbit.
  Interventions: Device: JOOL Health Mobile Phone Application

INTERVENTIONS:
Device: JOOL Health Mobile Phone Application — JOOL Health is a mobile phone-based application that aims to increase autonomous motivation to prevent T2DM by helping individuals make connections between certain health behaviors and the energy and willpower needed to achieve personal goals. On a daily basis, JOOL Health users chart the following health behaviors: Sleep, Presence, Activity, Creativity, and Eating. On a weekly basis, JOOL Health users are asked to record how well they lived according to their purpose and values. Through the integration of user-entered information with contextual data, JOOL Health provides tailored messaging and daily predictions of individuals' energy and willpower.
  Arms: JOOL-Only; JOOL-Plus

SUMMARY:
Type 2 diabetes mellitus (T2DM) can be prevented through weight loss and increased physical activity, yet its prevalence continues to rise. This trend may be due in part to low rates of participation in evidence-based lifestyle change programs such as the Diabetes Prevention Program (DPP). New strategies are needed to promote healthy behaviors among individuals at risk for T2DM, and mobile health technologies may be an effective and scalable approach to achieve this. One promising tool is JOOL Health, a mobile phone-based application that leverages principles from Self-Determination Theory to help individuals understand how certain behaviors (e.g. sleep, diet, physical activity) influence their ability to pursue their core values and purpose in life. Through personalized messaging and feedback, JOOL Health aims to increase autonomous motivation, a form of motivation closely associated with the initiation and maintenance of healthy behaviors.

In this mixed methods pilot randomized controlled trial, the investigators will test whether the JOOL Health mobile phone-based application -- used alone and in conjunction with other mobile health technologies to track weight and physical activity -- can increase autonomous motivation to prevent type 2 diabetes mellitus (T2DM) among individuals with prediabetes who previously declined participation in a Diabetes Prevention Program (DPP).

DETAILED DESCRIPTION:
This 12-week pilot randomized controlled trial aims to recruit 156 individuals with prediabetes who declined participation in a formal DPP despite invitation to participate at no out-of-pocket cost by their health plan. Participants will be randomized to 1 of 3 study arms: (1) a group that receives information on prediabetes, evidence-based strategies to decrease progression to diabetes, and a list of resources for mHealth tools for monitoring diet, physical activity, and weight (control group); (2) a group that receives the JOOL Health mobile phone application; and (3) a group that receives the JOOL Health mobile phone application and other mHealth tools (e.g. Fitbit activity tracker and wireless-enabled scale) whose results can be uploaded into JOOL.

The investigators will use a mixed methods approach with a sequential explanatory design, which is to say that quantitative data and qualitative data will be collected in 2 consecutive phases within the study. Specifically, in the first phase, investigators will collect and analyze qualitative data (e.g. focus groups) from a purposive sample of participants with differing levels of engagement and success. The rationale for this approach is that the quantitative data will provide a general overview of the intervention's efficacy and limitations, and the qualitative data will help to explain these findings by exploring participants' experiences and perspectives in more depth.

ELIGIBILITY:
Inclusion Criteria:

* Invited to participate in a DPP by the participant's health plan, but have not engaged in a program at least 6 months after receiving the first letter of invitation
* Wireless internet access
* Personal smartphone access

Exclusion Criteria:

* Individuals currently participating in another lifestyle or behavior change program or research study
* Inability to read, write, or speak English
* Inability to provide informed consent
* Women who are pregnant or intend to become pregnant during the intervention period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Autonomous Motivation to Prevent T2DM | 12 Weeks
  Change from baseline mean score on a scale of 1 - 7 as assessed by the Treatment Self Regulation Questionnaire- Autonomous Section survey instrument where 1 means little autonomous motivation and 7 means high autonomous motivation.

SECONDARY OUTCOMES:
Change in self-reported weight | Baseline to 12-week follow-up
Change in HbA1c | Baseline to 12-week follow-up
Change in psychosocial measures | Baseline to 12-week follow-up
  Overall motivation to prevent T2DM; purpose in life; perceived competence to prevent T2DM; social support; eating behavior; self-reported physical activity; patient activation; willingness to participate in a Diabetes Prevention Program

CONTACTS AND LOCATIONS:
Overall Officials: Dina Griauzde, MD, Study Director — Robert Wood Johnson Clinical Scholars Program (VA Scholar); Michele Heisler, MD, Principal Investigator — Robert Wood Johnson Clinical Scholars Program
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griauzde D, Kullgren JT, Liestenfeltz B, Ansari T, Johnson EH, Fedewa A, Saslow LR, Richardson C, Heisler M. A Mobile Phone-Based Program to Promote Healthy Behaviors Among Adults With Prediabetes Who Declined Participation in Free Diabetes Prevention Programs: Mixed-Methods Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 9;7(1):e11267. doi: 10.2196/11267. PMID 30626566
- [Derived] Griauzde DH, Kullgren JT, Liestenfeltz B, Richardson C, Heisler M. A mobile phone-based program to promote healthy behaviors among adults with prediabetes: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2018 Feb 13;4:48. doi: 10.1186/s40814-018-0246-z. eCollection 2018. PMID 29449958